CLINICAL TRIAL: NCT03899285
Title: Citalopram Titration in Early Non-responder Patients With Major Depressive Disorders: a Pilot Study (CRY-MOOD)
Brief Title: Citalopram Titration in Early Non-responder Patients With Major Depressive Disorders
Acronym: CRY-MOOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Marie-Claude Lefebvre, Principal investigator, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-1215
Record Dates: First submitted 2018-08-24; First posted 2019-04-02 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
Keywords: citalopram; major depressive disorder; non responder; MADRS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Preparation phase (Phase 1) : Every enrolled patients start with citalopram 10 mg daily for 3 days and 20 mg daily for 11 days.
  Escalation phase (Phase 2) :This phase is split in two arms which are the responders and the non-responders. Responders will pursue their citalopram 20 mg for 14 days. Non-responders will be assigned randomly 1:1 in 2 groups. Patients in group A will be randomized to receive a pill of citalopram 20 mg and a capsule of citalopram 20 mg for 14 days. The total dose of citalopram will be 40 mg once daily. Patients in group B receive a pill of citalopram 20 mg and a capsule of placebo (a capsule without medication) for 14 days. The total dose of citalopram will be 20 mg once daily.
  Follow-up phase (Phase 3) : Every responders will pursue their treatment of citalopram 20 mg daily for 28 days. It's possible that in this group, the treatment approach may vary depending the physician. Every non-responders (group A and B) will receive 40 mg of citalopram for 28 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Over-encapsulation was performed to maintain blind.
  Every participant will have the same step (visits, follow up, questionnaire and interview).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Citalopram increase (group A) (Experimental): At the end of the preparation phase, non-responders will be randomized to receive a pill of citalopram 20 mg and a capsule of citalopram 20 mg for a length of 14 days. The total dose of citalopram will be 40 mg once daily.
  Follow up will last 8 weeks in total.
  Interventions: Drug: Citalopram 20mg or 40 mg (phase 2)
- Placebo (group B) (Placebo Comparator): At the end of the preparation phase, non-responders will be randomized to receive a pill of citalopram 20 mg and a capsule of placebo (a capsule without medication) for a length of 14 days. The total dose of citalopram will be 20 mg once daily.
  Follow up will last 8 weeks in total.
  Interventions: Drug: Citalopram 20mg or 40 mg (phase 2)
- Observational arm (group c) (No Intervention): Eligible patients to this arm are responders to citalopram. A diminution of at least 30% of the symptoms from baseline with the MADRS is required to enter this arm. At the end of the first phase, these patients will pursue their citalopram 20 mg for the rest of the study (=6 weeks). It's possible that in this group, the treatment approach may vary depending the physician.
  Follow up will last 8 weeks in total.

INTERVENTIONS:
Drug: Citalopram 20mg or 40 mg (phase 2) — For non-responders, a randomisation 1:1 was chosen. The group A will receive 40 mg and the group B will receive 20 mg once daily of citalopram for 14 days.
  Arms: Citalopram increase (group A); Placebo (group B)

SUMMARY:
Major depressive disorder is a common mental disorder and the leading cause of disability worldwide. According to the Canadian Network for Mood and Anxiety Treatment, early improvement following an antidepressant treatment is correlated with response and remission. Escalation of an antidepressant dose after 2 weeks, as opposed to 4 to 8 weeks, is proposed to favor early improvement. However, this has never been tested systematically in a controlled study involving major depressive disorder patients that are non-responders to their antidepressant treatment.

DETAILED DESCRIPTION:
The investigators sought to assess whether it is feasible to perform a prospective randomized controlled double-blind feasibility study with a 2 week run-in period and 3 parallel groups randomized controlled study using citalopram. Citalopram has physicochemical properties compatible with over-encapsulation and a has a simple titration that allows the study of early dose increase.. It is among the most prescribed antidepressant in the province of Quebec and at the Hospital Maisonneuve-Rosemont - University family medicine group (U-FMG).

Since establishment of a randomized controlled trial is complex and expensive, a feasibility design is appropriate to identify all the obstacles and to minimize sources of possible bias (recruitment, follow up, resources).

ELIGIBILITY:
Inclusion Criteria:

* Understand french or english
* Primary diagnostic of major depressive disorder based on the Diagnostic and Statistical Manual of Mental Disorders criteria (5th edition)
* Prescription of citalopram
* Citalopram started less than 4 days ago
* Able to receive informed consent
* Not participating to another study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Unable to participate to follow-up
* Hypersensitivity to citalopram or any component of the formulation
* Known QT interval prolongation or congenital long QT syndrome
* Hepatic impairment (Child Pugh A, B or C)
* Renal impairment (Clcr < 30 ml/min)
* Known cytochrome P450 2C19 poor metabolizers
* History of non-response to citalopram
* Head trauma or severe cognitive impairment
* Substance-related and addictive disorders controlled less than 3 months or uncontrolled
* Schizophrenia or psychotic disorder
* Mixed depression
* History of manic/hypomanic episodes
* Use of prohibited drugs : monoamine oxidase inhibitors, cytochrome P450 2C19 inhibitors, drugs at risk of causing prolongation of the QT interval, cimetidine, pimozide and antidepressors taken for another psychiatric condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Primary outcomes determined by the proportion of non-responders (< 30 % improvement on the MADRS) after 2 weeks of treatment and the proportion of non-responders randomized patients who completed the study. | 8 weeks
  The efficacy of treatment was assessed by the Montgomery and Asberg Depression Rating Scale (MADRS).Threshold for non-responders : < 30 % improvement on the MADRS between T2 and T0. This scale was completed by a trained assessor and measures the severity of depressive episodes in patients with mood disorders. The scale is in french and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.
  Criteria for success of the randomization and completion of the study :
  * Sample size target : 24 non-responders randomized patients
  * Proportion of non-responders after 2 weeks of treatment (T2) : ≥ 0.45 (number of non-responders after 2 weeks of treatment divided by the number of enrolled patients).
  * Proportion of non-responders randomized patients who completed the full course of treatment (8 weeks) : ≥ 0.65 (number of non-responders randomized patients who completed the study divided by the total number of enrolled patients).

SECONDARY OUTCOMES:
Proportion of eligible subjects | 8 weeks
  Number of subjects who meet the eligibility criteria divided by the total number of patients referred to the study team.
Recruitment rate | 8 weeks
  Number of enrolled patients divided by total number of patients who meet the eligibility criteria.
Retention rate | 8 weeks
  Total number of patients who completed the full course of study divided by the number of enrolled patients.
  A descriptive analyse will be performed to identify the reasons of prematures departures.
Adherence rate to treatment | 8 weeks
  Assessed with pill count reported to the research pharmacy at each follow-up in clinic (T2, T4, T6 and T8).
Unblinding rate | 8 weeks
  Number of unblinded patients divided by the total number of enrolled patients.
  A descriptive analyse will be performed to identify the reasons of unblinding.
Length of interviews | 8 weeks
  An average of all the interviews will be calculated (in minutes).
Side effects reported to the assessors and measured by the Frequency, Intensity, and Burden of Side Effect Rating (FIBSER). | 8 weeks
  The side effects were reported to assessor and their gravity were measured by a self-administrated scale called the FIBSER.The FIBSER is composed of 3 questions and takes 3 distinct aspects : frequency, intensity and the burden of side effect on the quality of life. The scale was in french and has 3 questions, with an overall score ranging from 0 to 18 points. Higher score indicates a high side-effect burden that should be evaluated.
Response curves for all patients according to the results from the MADRS. | 8 weeks
  Compare the clinical response following the increase of citalopram at 2 weeks (group A) or 4 weeks (group B) in non-responder patients according to the results from the Montgomery and Asberg Depression Rating Scale (MADRS) at T2, T4, T6 and T8.
  This scale was completed by a trained assessor and measures the severity of depressive episodes in patients with mood disorders. The scale is in french and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.
Correlation between the results of Patient Health Questionnaire-9 (PHQ-9) and the MADRS at each follow-up (T2, T4, T6 and T8). | 8 weeks
  A pearson coefficient to describe the correlation (r) between the PHQ-9 and the Montgomery and Asberg Depression Rating Scale (MADRS) was chosen.
  The PHQ-9 is a questionnaire self-reported assessing the severity of the depression. The scale was in french and has 9 items, with an overall score ranging from 0 to 27 points. Higher score indicates more severe depression.
  The MADRS was completed by a trained assessor and measures the severity of depressive episodes in patients with mood disorders. The scale is in french and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Lefebvre, MD, Principal Investigator — GMF-U Maisonneuve-Rosemont Hospital
Locations (1):
- GMF-U Maisonneuve-Rosemont hospital, Montreal East, Quebec, Canada